CLINICAL TRIAL: NCT06480032
Title: Low-Load Blood Flow Restriction Training vs Traditional Resistance Training Exercises Following Anterior Cruciate Ligament Reconstruction Surgery: A Pilot Randomized Controlled Trial
Brief Title: Low-Load Blood Flow Restriction Training vs Traditional Resistance Training Exercises Following ACLR Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abasyn University Peshawar (Other)
Collaborators: Nazarbayev University (Other)
Responsible Party: Principal Investigator, Mohammad Shoaib khan, Doctor, Abasyn University Peshawar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AbasynU
Record Dates: First submitted 2024-04-15; First posted 2024-06-28 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Strength; Range of Motion; Pain-Knee; Skeletal Muscle Hypertrophy; Effusion Joint
Keywords: Blood Flow Restriction Training; Resistance Training; Anterior Cruciate Ligament Reconstruction; Skeletal Muscle Hypertrophy
MeSH Terms: conditions — Hydrarthrosis

STUDY DESIGN:
Intervention Model Description: BFR with standard post-operative rehabilitation for 8 weeks followed by the standard protocol progression for the remainder of the treatment program. The other group (Group 2) receive standard post-operative rehabilitation without BFR for the duration of treatment program.
Who Masked: Investigator
Masking Description: Single-assessor blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blood Flow Restriction band (Experimental): Group 1, comprising 16 patients (Group 1), undergo the standard Anterior Cruciate Ligament (ACL) rehabilitation protocol with Blood Flow Restriction (BFR) for 8 weeks during their physiotherapy sessions at the Rehman Medical Institute's Outpatient Department (OPD), starting from the second post-operative visit. The cuff size determined based on the patient's thigh circumference.
  The rehabilitation protocol will progress as follows:
  * Week 2-4: Long Arc Quadriceps (LAQ) exercise progression, Shuttle exercise progression, and Post-op visit 2.
  * Week 4-8: Available range LAQ, Standing terminal knee extension, and Single Limb Shuttle/Leg Press exercises.
  Interventions: Device: Blood Flow Restriction band
- Non-Blood Flow Restriction band (Other): Group B, comprising 16 patients (Group 2), undergo the standard Anterior Cruciate Ligament (ACL) rehabilitation protocol without Blood Flow Restriction (BFR) for 8 weeks during their physiotherapy sessions at the Rehman Medical Institute's Outpatient Department (OPD), starting from the second post-operative visit. The cuff size determined based on the patient's thigh circumference.
  The rehabilitation protocol will progress as follows:
  * Week 2-4: Long Arc Quadriceps (LAQ) exercise progression, Shuttle exercise progression, and Post-op visit 2.
  * Week 4-8: Available range LAQ, Standing terminal knee extension, and Single Limb Shuttle/Leg Press exercises.
  Interventions: Device: Blood Flow Restriction band

INTERVENTIONS:
Device: Blood Flow Restriction band — Blood Flow Restriction (BFR) band operate by partially occluding arterial blood flow to distal structures, but more significantly impeding venous outflow from under the cuff, thereby also hindering venous return. The compression of vasculature proximal to the skeletal muscle leads to inadequate oxygen supply (hypoxia) within the muscle tissue, resulting in a localized hypoxic environment. Additionally, the reduction in venous blood flow causes blood to accumulate in the capillaries of the occluded limb, often manifesting as visible erythema. This temporary restriction will be maintained for a duration of 8 weeks.
  Other Names: Brand name: Fitbiz Exercise Equipment

SUMMARY:
The main objective/s of the study is to compare the effectiveness of low load blood flow restriction training (LL-BFR) with traditional resistance training exercises (T-RT) at improving skeletal muscle hypertrophy, strength, Range of motion (ROM), pain and effusion in individuals who have undergone anterior cruciate ligament (ACL) reconstruction surgery.

The study involves 32 participants who meet the inclusion criteria and randomly assign to either BFR-RT group or the T-RT group. The primary outcomes measured includes skeletal muscle hypertrophy, strength, range of motion, pain, and effusion.

The intervention last for eight weeks, during which participants undergone resistance training according to their assigned group. Data collected at various time points, including post-surgery, mid-training, and post-training, to assess the effectiveness of the two training methods. The findings from this study are effective for anterior cruciate ligament reconstruction surgery (ACLR) patients in early rehabilitation and improve outcomes for individuals recovering from ACL injuries.

DETAILED DESCRIPTION:
The purpose of this randomized controlled trial is to compare the effectiveness of low-load blood flow restriction training (BFR-RT) with low-load traditional resistance training exercises (T-RT) in individuals who have undergone anterior cruciate ligament reconstruction (ACLR) surgery. The anterior cruciate ligament is a major knee ligament that provides stability to the knee joint. ACL injuries are common, and surgical reconstruction is often necessary to restore knee stability and function.

The study was conducted at Rehman Medical Institute over approximately one and a half years. The sample size consists of 32 participants who meet the inclusion criteria, including having undergone unilateral ACLR surgery within the past 8 weeks and being free of any neurological impairments or significant cardiac, pulmonary, or metabolic conditions.

Participants were randomly assigned to either the BFR-RT or T-RT group using a random sampling technique. Randomization was conducted by an independent member of the research team using opaque envelopes containing coded group assignments to ensure unbiased allocation.

The intervention involved 8 weeks of biweekly unilateral leg training on the affected limb under the instruction of a physiotherapist, totaling 16 training sessions. Participants in both groups received the standard rehabilitation program provided by the hospital. In the BFR-RT group, blood flow restriction was achieved using an occlusion band placed on the most proximal portion of the affected limb. The physical therapist ensured the band was not too tight, allowing one finger to pass through the band.

Data were collected at three time points: post-surgery (week 0-1), mid-training (week 4-5), and post-training (week 9). Outcomes measured included skeletal muscle hypertrophy, strength (assessed using manual muscle testing), range of motion (ROM) of the knee joint, pain (assessed using a Knee Injury and Osteoarthritis Outcome Score), and effusion (measured by knee joint circumference). Adherence rates, exercise session attendance, and no adverse events were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Post-ACL reconstruction surgery (week 0-8)
* Both male and female
* No known history of central or peripheral neurological impairment
* Free of any cardiac, pulmonary or metabolic conditions
* Willing to participate

Exclusion Criteria:

* History of deep vein thrombosis or vascular pathology in any lower limb
* Intraarticular injections into the knee in the preceding 6 months
* Rheumatoid arthritis or other significant co-morbidities
* Use of anticoagulant medications

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-06-04 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Khan, Master's, Study Chair — Rehman Medical Institute
Locations (1):
- Rehman Medical Institute, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
IPD will be share during and after the study completion with other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: Within a 1-year timeframe, the study will share all required documents and SAPs with other researchers.
Access Criteria: PDF

REFERENCES:
- [Background] Scott BR, Loenneke JP, Slattery KM, Dascombe BJ. Exercise with blood flow restriction: an updated evidence-based approach for enhanced muscular development. Sports Med. 2015 Mar;45(3):313-25. doi: 10.1007/s40279-014-0288-1. PMID 25430600
- [Background] Sanders TL, Maradit Kremers H, Bryan AJ, Larson DR, Dahm DL, Levy BA, Stuart MJ, Krych AJ. Incidence of Anterior Cruciate Ligament Tears and Reconstruction: A 21-Year Population-Based Study. Am J Sports Med. 2016 Jun;44(6):1502-7. doi: 10.1177/0363546516629944. Epub 2016 Feb 26. PMID 26920430
- [Background] Khalid K, Anwar N, Saqulain G, Afzal MF. Neuromuscular Training following Anterior Cruciate Ligament reconstruction - Pain, Function, Strength, Power & Quality of Life Perspective: A Randomized Control Trial. Pak J Med Sci. 2022 Nov-Dec;38(8):2175-2181. doi: 10.12669/pjms.38.8.5730. PMID 36415269

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical hospital
Pre-assignment Details: There were no excluded participants of enrolled groups during data collection.
Groups:
- Non-Blood Flow Restriction Band: Group B, comprising 16 patients (Group 2), undergo the standard Anterior Cruciate Ligament (ACL) rehabilitation protocol without Blood Flow Restriction (BFR) for 8 weeks during their physiotherapy sessions at the Rehman Medical Institute's Outpatient Department (OPD), starting from the second post-operative visit. The cuff size determined based on the patient's thigh circumference.
  The rehabilitation protocol will progress as follows:
  * Week 2-4: Long Arc Quadriceps (LAQ) exercise progression, Shuttle exercise progression, and Post-op visit 2.
  * Week 4-8: Available range LAQ, Standing terminal knee extension, and Single Limb Shuttle/Leg Press exercises.
  Blood Flow Restriction band: Blood Flow Restriction (BFR) band operate by partially occluding arterial blood flow to distal structures, but more significantly impeding venous outflow from under the cuff, thereby also hindering venous return. The compression of vasculature proximal to the skeletal muscle leads to inadequate oxygen supply (hypoxia) within the muscle tissue, resulting in a localized hypoxic environment. Additionally, the reduction in venous blood flow causes blood to accumulate in the capillaries of the occluded limb, often manifesting as visible erythema. This temporary restriction will be maintained for a duration of 8 weeks.
- Blood Flow Restriction Band: Group 1, comprising 16 patients (Group 1), undergo the standard Anterior Cruciate Ligament (ACL) rehabilitation protocol with Blood Flow Restriction (BFR) for 8 weeks during their physiotherapy sessions at the Rehman Medical Institute's Outpatient Department (OPD), starting from the second post-operative visit. The cuff size determined based on the patient's thigh circumference.
  The rehabilitation protocol will progress as follows:
  * Week 2-4: Long Arc Quadriceps (LAQ) exercise progression, Shuttle exercise progression, and Post-op visit 2.
  * Week 4-8: Available range LAQ, Standing terminal knee extension, and Single Limb Shuttle/Leg Press exercises.
  Blood Flow Restriction band: Blood Flow Restriction (BFR) band operate by partially occluding arterial blood flow to distal structures, but more significantly impeding venous outflow from under the cuff, thereby also hindering venous return. The compression of vasculature proximal to the skeletal muscle leads to inadequate oxygen supply (hypoxia) within the muscle tissue, resulting in a localized hypoxic environment. Additionally, the reduction in venous blood flow causes blood to accumulate in the capillaries of the occluded limb, often manifesting as visible erythema. This temporary restriction will be maintained for a duration of 8 weeks.
Period: Overall Study
Arm/Group | Non-Blood Flow Restriction Band | Blood Flow Restriction Band
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data were analyzed by checking the normality of data. Sample T test and Mann Whitney U test were used for two groups
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Blood Flow Restriction Band | Blood Flow Restriction Band | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 11 | 14 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Pakistan | 16 | 16 | 32
Region of Enrollment [Number; unit: participants]
  Pakistan | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Range of Motion
Description: Knee range of motion assessed weekly for eight consecutive weeks with the patient in a supine position using goniometer.
Time Frame: eight weeks
Measure: Mean (Standard Deviation); unit: Degrees
Groups:
- Blood Flow Restriction Band: Group 1, comprising 16 patients (Group 1), undergo the standard Anterior Cruciate Ligament (ACL) rehabilitation protocol with Blood Flow Restriction (BFR) for 8 weeks during their physiotherapy sessions at the Rehman Medical Institute's Outpatient Department (OPD), starting from the second post-operative visit.
  The rehabilitation protocol will progress as follows:
  * Week 2-4: Long Arc Quadriceps (LAQ) exercise progression, Shuttle exercise progression, and Post-op visit 2.
  * Week 4-8: Available range LAQ, Standing terminal knee extension, and Single Limb Shuttle/Leg Press exercises.
  Blood Flow Restriction band: Blood Flow Restriction (BFR) band operate by partially occluding arterial blood flow to distal structures, but more significantly impeding venous outflow from under the cuff, thereby also hindering venous return. The compression of vasculature proximal to the skeletal muscle leads to inadequate oxygen supply (hypoxia) within the muscle tissue, resulting in a localized hypoxic environment.
Arm/Group | Blood Flow Restriction Band | Non-Blood Flow Restriction Band
Number analyzed (Participants) | 16 | 16
Degrees | 74.0625 (14.04976) | 80.3125 (14.65933)

2. Primary Outcome: Quadricep Strength
Description: Strength assessed through manual muscle testing (MMT). The grading scale ranges from 0 to 5, with Grade 0 indicating no visible or palpable muscle contraction and Grade 5 indicates muscle movement against gravity and maximal resistance.
Time Frame: eight weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Blood Flow Restriction Band: Group 1, comprising 16 patients (Group 1), undergo the standard Anterior Cruciate Ligament (ACL) rehabilitation protocol with Blood Flow Restriction (BFR) for 8 weeks during their physiotherapy sessions at the Rehman Medical Institute's Outpatient Department (OPD), starting from the second post-operative visit. The cuff size determined based on the patient's thigh circumference.
  Muscle strength was analyzed as follows:
  Quadriceps strength was assessed with the patient in a supine lying position during the first and second weeks following anterior cruciate ligament reconstruction surgery.
  In the fourth to sixth week, muscle strength were analyzed while the patients were in a seated position, with the leg hanging freely to allow resistance to be applied against the physiotherapist's hand.
- Non-Blood Flow Restriction Band: Group B, comprising 16 patients (Group 2), undergo the standard Anterior Cruciate Ligament (ACL) rehabilitation protocol without Blood Flow Restriction (BFR) for 8 weeks during their physiotherapy sessions at the Rehman Medical Institute's Outpatient Department (OPD), starting from the second post-operative visit.
  Muscle strength was analyzed as follows:
  Quadriceps strength was assessed with the patient in a supine lying position during the first and second weeks following anterior cruciate ligament reconstruction surgery.
  In the fourth to sixth week, muscle strength were analyzed while the patients were in a seated position, with the leg hanging freely to allow resistance to be applied against the physiotherapist's hand.
Arm/Group | Blood Flow Restriction Band | Non-Blood Flow Restriction Band
Number analyzed (Participants) | 16 | 16
units on a scale | 3.9375 (3.5) | .6800735 (.5163978)

3. Primary Outcome: Knee Pain
Description: Pain was assessed using visual analogue scale. This questionnaire ranges 0 to 10, where 10 indicates the worst pain and 0 indicates no pain. A higher score reflects higher pain.
Time Frame: eight weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Blood Flow Restriction Band; Non-Blood Flow Restriction Band: Group 1, muscle strength was analyzed as follows:
  Pain was assessed using a visual analogue scale (VAS) questionnaire at three different intervals: post-surgery, mid-training, and post-training.
Arm/Group | Blood Flow Restriction Band | Non-Blood Flow Restriction Band
Number analyzed (Participants) | 16 | 16
units on a scale | 2.0625 (1.12361) | 1.9375 (1.340087)

4. Primary Outcome: Quadricep Size
Description: Muscle size assessed using measuring tap wrapping around the thigh of pre-patellar region.
Time Frame: eight weeks
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Blood Flow Restriction Band: Muscle size were analyzed using measuring tape to measure the diameter the thigh of proximal patellar region
- Non-Blood Flow Restriction Band: Muscle size were analyzed using measuring tape to measure the diameter the thigh of proximal patellar region in three different occasions; post surgery, mid surgery and post training.
Arm/Group | Blood Flow Restriction Band | Non-Blood Flow Restriction Band
Number analyzed (Participants) | 16 | 16
cm | 19.375 (2.028957) | 18.65625 (2.650275)

ADVERSE EVENTS:
Time Frame: Adverse effects were not assessed.
Description: Adverse effects were not monitored.
Groups:
- Blood Flow Restriction Band; Non-Blood Flow Restriction Band: Adverse effects were not assessed
Arm/Group | Blood Flow Restriction Band | Non-Blood Flow Restriction Band
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Sample size was small

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT06480032/Prot_SAP_000.pdf